CLINICAL TRIAL: NCT07276269
Title: Comparative Study of Survival and Success of Restorations Exclusively Using the CAD/CAM Digital Method After 5 Years of Intraoral Use
Brief Title: Survival and Success of CAD/CAM Restorations After 5 Years of Intraoral Use
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 157/04-04-2022
Record Dates: First submitted 2025-04-02; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Tooth Wear
Keywords: CAD/CAM; Lithium Disilicate; Digital Dentistry
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAD/CAM Restoration Arm (Experimental): This arm involves the placement of dental restorations using CAD/CAM technology. Participants receive restorations fabricated through a digital workflow, which includes intraoral scanning, CAD software design, and milling of the restorations using CAM equipment. The restorations are made from high-quality ceramic or composite materials, chosen based on their suitability for long-term intraoral use. The process eliminates the need for conventional impression techniques, ensuring a precise fit. Participants are monitored over a 5-year period to evaluate the survival rate and success of the restorations, focusing on factors such as marginal integrity, wear resistance, and patient-reported outcomes.
  Interventions: Device: CAD/CAM Digital Restoration Placement; Device: Study of the Survival and Success of Endodontic Posts Using the CAD/CAM Digital Method After 5 Years of Intraoral Use

INTERVENTIONS:
Device: CAD/CAM Digital Restoration Placement — This intervention involves the placement of dental restorations exclusively using CAD/CAM technology, which includes digital scanning, design, and milling of the restorations. The restorations are fabricated from high-quality ceramic or composite materials that are commonly used in CAD/CAM systems. The process begins with an intraoral scan to capture the patient's dental anatomy, followed by the design of the restoration using CAD software, and milling with CAM equipment. The restorations are then adjusted, finished, and cemented intraorally. This intervention is distinct as it utilizes a fully digital workflow without the use of conventional impression techniques, aiming to assess the long-term clinical performance, survival rate, and success of these restorations over a period of 5 years. The study monitors factors such as restoration integrity, marginal adaptation, wear resistance, and patient-reported outcomes
  Other Names: Digital Dental Restoration; Intraoral Scanning Technique
Device: Study of the Survival and Success of Endodontic Posts Using the CAD/CAM Digital Method After 5 Years of Intraoral Use — This intervention involves the exclusive use of the CAD/CAM digital method for fabricating and placing endodontic posts. The study evaluates the long-term survival and success rate of these posts over a period of 5 years in an intraoral setting. This method is distinct as it eliminates the need for traditional impression techniques, utilizing digital scanning and milling for precise and consistent post fabrication. The focus is on comparing outcomes with those of conventional analog methods to establish the efficacy and reliability of the CAD/CAM approach.

SUMMARY:
This study evaluates the survival and success rates of dental restorations fabricated exclusively using CAD/CAM technology over a period of 5 years. The study will involve placing CAD/CAM restorations using a digital workflow that includes intraoral scanning, computer-aided design (CAD), and computer-aided manufacturing (CAM). The restorations will be monitored for factors such as marginal adaptation, wear resistance, and patient-reported outcomes. The goal is to determine the long-term clinical effectiveness of CAD/CAM restorations compared to traditional methods. The findings aim to improve the understanding and application of digital dental technology in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Patients with single or multiple CAD/CAM restorations placed within the last 5 years
* Adequate oral hygiene and willingness to participate in follow-up assessments
* Healthy periodontal status or controlled periodontal condition Signed informed consent form

Exclusion Criteria:

* Patients with systemic diseases affecting oral health (e.g., diabetes, osteoporosis)
* Pregnant or breastfeeding individuals
* Smokers or individuals with a history of heavy smoking
* Patients with untreated dental caries or advanced periodontal disease
* Individuals with previous allergic reactions to CAD/CAM materials used

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Survival Rate of CAD/CAM Restorations Over 5 Years | 5 years post-restoration
  This outcome measure evaluates the survival rate of CAD/CAM restorations over a 5-year period. Survival is defined as restorations remaining functional without failure such as fracture, debonding, or significant wear that would require replacement or major repair."

CONTACTS AND LOCATIONS:
Overall Officials: KOSMAS TOLIDIS, PROFESSOR, Study Chair — PROFESSOR, SCHOOL OF DENTISTRY, ARISTOTLE UNIVERISTY OF THESSALONIKI
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece